CLINICAL TRIAL: NCT04282161
Title: Pivotal Study of the Medtronic Axys EX Rotational Atherectomy System for the Treatment of Peripheral Arterial Disease in the Vasculature of the Lower Limbs
Brief Title: Pivotal Study of the Medtronic Axys EX Rotational Atherectomy System
Acronym: Axys ACHIEVE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT17045
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Vascular Disease; Critical Limb Ischemia; Superficial Femoral Artery Stenosis; Atherosclerosis; Arteriosclerosis; Vascular Diseases; Arterial Disease Occlusive; lower extremity arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia; Atherosclerosis; Arteriosclerosis; Vascular Diseases; Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Axys EX device (Experimental)
  Interventions: Device: Axys EX device

INTERVENTIONS:
Device: Axys EX device — Rotational atherectomy system for endovascular treatment of peripheral arterial disease prior to adjunctive therapy, if needed
  Other Names: Axys EX

SUMMARY:
The primary objective is to demonstrate the safety and effectiveness of the Axys EX rotational atherectomy system in subjects with peripheral arterial disease who have de novo or non-stented restenotic obstructive lesions in the peripheral vasculature of the lower limbs.

ELIGIBILITY:
General Inclusion Criteria:

1. Rutherford Clinical Category (RCC) Score of 2 - 5
2. Willing and capable of complying with all follow-up evaluations at the specified times
3. Age ≥ 18 years old
4. Provides written informed consent prior to study specific procedures
5. Completed Ankle/Brachial Index (ABI) (or Toe/Brachial Index [TBI]) prior to index procedure (up to 60 days prior)

   Angiographic Inclusion Criteria:
6. Evidence of ≥ 70% stenosis or occlusion in the peripheral vasculature of the target vessel, confirmed by angiography
7. Target lesion present in a single limb that consists of a single de novo or non-stented restenotic lesion, or qualifies as a tandem or combination lesion per the definitions below:

   1. Tandem (adjacent) Lesion: Lesions present in the same target vessel that can be treated as one single lesion and is separated by an angiographic normal vessel ≤3 cm at any point. Multiple points of separation can be present in single lesion treatment if no single point of separation is > 3 cm
   2. Combination Lesion: A single lesion that is not completely occluded but includes a segment of complete occlusion anywhere along the length
8. Exchangeable guidewire must cross target lesion within the lumen
9. Total target lesion length is ≥ 20 mm and ≤ 200mm
10. Reference vessel diameter (RVD) is ≥ 2.0 mm and ≤ 5.0 mm
11. Identifiable distal target vessel which upon completion of the intervention is anticipated to provide reconstitution of blood flow to the foot. Angiographic evidence of adequate distal runoff through the foot (at least one native calf vessel [posterior tibial, anterior tibial, or peroneal artery] is patent, defined as < 50% stenosed)
12. Multiple lesions in the target limb (including the target lesion and non-target lesions) may be treated if all of the following applies:

    1. Non-target lesion(s) must be located proximal to the target lesion
    2. Non-target lesion(s) must be successfully treated (defined as optimally treated [e.g. no untreated arterial dissections or perforation present]) by standard endovascular procedures prior to initiation of treatment of the target lesion
    3. Non-target lesions treated prior to target lesion cannot be treated with rotational, orbital or laser atherectomy
    4. Non-target lesion(s) may be located in separate vascular beds (i.e., iliac,femoropopliteal, tibial) or multiple tibial vascular beds (i.e., anterior tibial, posterior tibial, tibioperoneal trunk/peroneal). (Note: Only one tibial vessel may be identified as the target vessel with the target lesion.)
    5. Only one lesion per the above definitions may be treated as the target lesion with the Axys EX device

    General Exclusion Criteria:
13. Has one or more of the contraindications listed in the Axys EX Rotational Atherectomy System's IFU
14. Contraindication or known untreated allergy to antiplatelet therapy, anticoagulants, thrombolytic drugs, or any other drug anticipated to be used
15. Hypersensitivity to contrast material that cannot be adequately pretreated
16. Known uncontrollable hypercoagulable condition or refuses blood transfusion
17. Life expectancy of less than 12 months
18. Surgical (requiring hospitalization) or endovascular intervention of the target limb within 30 days prior to the index procedure
19. Planned surgical intervention or endovascular procedure within 30 days after the index procedure
20. Currently participating in an investigational drug or another device study that may clinically interfere with the study endpoints
21. Other co-morbid condition(s) that in the judgment of the physician precludes safe percutaneous intervention
22. If a previous peripheral bypass affecting the target limb is present, the bypass must be patent and the target lesion cannot be present in the peripheral bypass artery
23. Impaired renal function (defined as GFR < 30 mL/min) or on dialysis
24. Recent myocardial infarction or stroke ≤ 30 days prior to the index procedure
25. Previous or planned amputation above the metatarsal line on the target limb
26. Patient belongs to a vulnerable population per investigator's judgment or patient has any kind of disorder that compromises his/her ability to give written informed consent and/or to comply with study procedures. Patient must be able to consent for themselves
27. Patient is pregnant (female patients of child-bearing potential must have a pregnancy test done within 7 days prior to the index procedure)

    Angiographic Exclusion Criteria:
28. Noted thrombus at the point of the intended target lesion
29. In-stent restenosis of the target lesion
30. Aneurysmal target vessel
31. Hemodynamic significant stenosis or occlusion of inflow tract that has not been revascularized prior to treatment of the target vessel
32. Perforation, flow limiting dissection or other injury of the target vessel requiring surgical intervention prior to enrollment
33. Disease that precludes safe advancement of the Axys EX device to the target lesion
34. Need to treat a lesion distal to the target index lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness | During procedure
  Change in percent stenosis in the treatment vessel. Percent stenosis is defined as native vessel diameter as measured at the narrowest point of the lesion divided by the estimated native vessel diameter at that location.
Primary Safety | 30-Days
  Major Adverse Events (MAEs) at 30 Days post-procedure defined as freedom from clinically-driven target lesion revascularization (CD-TLR), major unplanned amputation of the treated limb, or all-cause mortality.

SECONDARY OUTCOMES:
Technical Success | During Procedure
  Defined as the ability of the Axys EX device to successfully traverse/cross the entire intended length of the target lesion
Procedural Success | During Procedure
  Defined as ≤ 30% residual stenosis following use of the Axys EX device and adjunctive therapy as measured by angiography and determined by the angiographic core laboratory
Amputation-Free Survival | 12-Months
  Defined as freedom from a major, unplanned amputation of the target limb through the 12 month visit
Major Adverse Events (MAEs) | 12-Months
  Defined as freedom from clinically-driven target vessel revascularization (CD-TVR), major unplanned amputation of the treated limb, thrombosis at the target lesion site, or all-cause mortality
Rate of Target Lesion Revascularization (TLR) | 6 and 12-Months
  Any re-intervention at the target lesion
Rate of Target Vessel Revascularization (TVR) | 6 and 12-Months
  Any re-intervention within the target vessel
Provisional Stent Rate | During Procedure
Flow Limiting Dissection | During Procedure
  Target lesion flow limiting dissection (D or greater) rate after adjunctive therapy
Primary Patency as determined by Duplex Ultrasound (DUS) | 6 and 12-Months
  1. For subjects with a target lesion in the femoropopliteal region (above the knee [ATK]) through the level of popliteal segment P3 (below the knee popliteal artery from the center of the knee joint space to the origin of anterior tibial artery), primary patency is defined as freedom from core laboratory-assessed restenosis (DUS PSVR ≤2.4) and CD-TLR (adjudicated by a Clinical Events Committee)
  2. For subjects with a target lesion below the level of popliteal segment P3 (below the knee [BTK]), primary patency is defined as freedom from core laboratory-assessed absence of target lesion occlusion (no flow) as assessed by DUS and CD-TLR (adjudicated by a Clinical Events Committee)
Quality of Life Assessment | 30-Days, 6 and 12-Months
  EQ-5D questionnaire
Walking Distance | 30-Days, 6 and 12-Months
  6-Minute Walking Test
Walking Capacity | 30-Days, 6 and 12-Months
  Walking Impairment Questionnaire (WIQ)
Ankle/brachial index (ABI) or toe/brachial index (TBI) | 30-Days, 6 and 12-Months
Rutherford clinical category (RCC) | 30-Days, 6 and 12-Months
Distal Embolization in Target Limb | 30-Days
  Clinically significant distal embolization in target limb within 30 days defined as distal embolization requiring treatment by mechanical or pharmacologic means (other than a vasodilator) (adjudicated by a Clinical Events Committee)
Major Vessel Perforation | 30-Days
  requiring surgical or endovascular repair within 30 days (adjudicated by a Clinical Events Committee) 6.

CONTACTS AND LOCATIONS:
Overall Officials: Ravish Sachar, MD FACC, Principal Investigator — North Carolina Heart and Vascular; Brian DeRubertis, MD FACS, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No